CLINICAL TRIAL: NCT02489045
Title: Noninvasive Subharmonic Aided Pressure Estimation of Portal Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: University of Pennsylvania (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14F.113; R01DK098526 (NIH)
Record Dates: First submitted 2015-05-14; First posted 2015-07-02 (Estimated); Results first posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-07

CONDITIONS: Liver Diseases; Portal Hypertension
MeSH Terms: conditions — Liver Diseases; Hypertension, Portal | interventions — Sonazoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SHAPE measurement (Experimental): 48 µl of Sonazoid microbubbles (GE Healthcare, Oslo, Norway) will be co-infused at a rate of 0.024 µl/kg body weight/minute together with a 0.9% NaCl solution infused at a rate of at least 2 ml/min.
  Interventions: Drug: SHAPE measurement (Sonazoid ultrasoud contrast agent)

INTERVENTIONS:
Drug: SHAPE measurement (Sonazoid ultrasoud contrast agent) — Three vials with 48 µl of Sonazoid (GE Healthcare, Oslo, Norway) microbubbles (6 ml) will be prepared and drawn into a 10 ml syringe, placed in a syringe pump. Sonazoid will be co-infused at a rate of 0.024 µl/kg body weight/minute (suspension infusion rate of 0.18 ml/kg/hour) together with a 0.9% NaCl solution infused at a rate of at least 2 ml/min.
  Other Names: Sonazoid

SUMMARY:
This is an open-label, non-randomized trial that will be conducted at two clinical sites, Thomas Jefferson University (TJU) and the Hospital of the University of Pennsylvania (HUP). Enrolled patients undergoing trans-jugular liver biopsy with hepatic vein pressure gradient (HVPG) measurements will receive a continuous infusion of Sonazoid® (GE Healthcare, Oslo, Norway) co-infused with 0.9% NaCl solution over a 5-10 minute time period. Ultrasound imaging will be performed using a Logiq 9 scanner with a 4C transducer (GE Healthcare, Milwaukee, WI) and the novel SHAPE (subharmonic aided pressure estimation) algorithm will be used to measure pressure values in the hepatic and portal veins. Data will be stored on a PC and compared to pressure-catheter measurements, Subjects identified in the initial examination as having portal hypertension (by HVPG results) will be monitored by SHAPE for up to 18 months. These subjects typically have surveillance Computed tomography (CT) or magnetic resonance imaging (MRI) scans every 6 months to screen for liver cancer, and at those times a repeat SHAPE examination will be performed (ideally within 1 month of their clinically indicated imaging follow up appointment). In patients who undergo more frequent screening (generally 3 month intervals), SHAPE exams will be performed at 6 month intervals. Any repeat trans-jugular liver biopsies performed in this population will also trigger a repeat SHAPE study. Results of blood test evaluations (performed every 3 months in this population), medication, concomitant imaging study or procedure (including endoscopies) will be noted (all blood tests and imaging are clinically indicated only and are not required by this protocol). The end point for this part of the study will be any one new complication (e.g., liver cancer) or a marked worsening in any complication, liver transplantation, death, or the end of this clinical trial (after 3 years). The investigators expect these patients will be monitored three times during the course of this clinical trial. The time to reach the end point will be noted if a new complication or a marked worsening in any complication occurs.

ELIGIBILITY:
Inclusion Criteria:

* Be scheduled for trans-jugular liver biopsy the day of the ultrasound procedure.
* Be at least 21 years of age.
* Be medically stable.
* If a female of child-bearing potential, must have a negative pregnancy test.
* Be conscious and able to comply with study procedures.
* Have read and signed the IRB-approved Informed Consent form for participating in the study.

Exclusion Criteria:

* Females who are pregnant or nursing.
* Patients not scheduled for trans-jugular liver biopsy
* Patients who have received an investigational drug in the 30 days before study drug administration, or will receive one within 72 h afterwards,.
* Patients with known or suspected right-to-left, bi-directional, or transient right-to-left cardiac shunts
* Patients with pulmonary hypertension or unstable cardiopulmonary conditions
* Patients currently on chemotherapy or with other primary cancers requiring systemic or hepatic loco-regional treatment.
* Patients who are medically unstable, patients who are seriously or terminally ill, and patients whose clinical course is unpredictable. For example:
* Patients on life support or in a critical care unit.
* Patients with unstable occlusive disease (e.g., crescendo angina)
* Patients with clinically unstable cardiac arrhythmias, such as recurrent ventricular tachycardia.
* Patients with uncontrolled congestive heart failure (NYHA Class IV)
* Patients with recent cerebral hemorrhage.
* Patients who have undergone surgery within 24 hours prior to the study sonographic examination.
* Patients with a history of anaphylactic allergy to eggs or egg products, manifested by one or more of the following symptoms: generalized urticaria, difficulty in breathing, swelling of the mouth and throat, hypotension, or shock. (Subjects with nonanaphylactic allergies to eggs or egg products may be enrolled in the study, but must be watched carefully for 1 h following the administration of SONAZOID).
* Patients with congenital heart defects.
* Patients with severe emphysema, pulmonary vasculitis, or a history of pulmonary emboli.
* Patients with respiratory distress syndrome
* Patients with thrombosis within the hepatic, portal, or mesenteric veins.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2015-04-06 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flemming Forsberg, PhD, Principal Investigator — Thomas Jefferson University
Locations (2):
- United States (2):
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Dept of Radiology, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Eisenbrey JR, Dave JK, Halldorsdottir VG, Merton DA, Miller C, Gonzalez JM, Machado P, Park S, Dianis S, Chalek CL, Kim CE, Baliff JP, Thomenius KE, Brown DB, Navarro V, Forsberg F. Chronic liver disease: noninvasive subharmonic aided pressure estimation of hepatic venous pressure gradient. Radiology. 2013 Aug;268(2):581-8. doi: 10.1148/radiol.13121769. Epub 2013 Mar 22. PMID 23525208
- [Derived] Gupta I, Eisenbrey JR, Machado P, Stanczak M, Wessner CE, Shaw CM, Gummadi S, Fenkel JM, Tan A, Miller C, Parent J, Schultz S, Soulen MC, Sehgal CM, Wallace K, Forsberg F. Diagnosing Portal Hypertension with Noninvasive Subharmonic Pressure Estimates from a US Contrast Agent. Radiology. 2021 Jan;298(1):104-111. doi: 10.1148/radiol.2020202677. Epub 2020 Nov 17. PMID 33201789

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SHAPE Measurement
Started | 178
Completed | 125
Not Completed | 53
Not completed — unable to collect usable data | 53
Period: Follow-up
Arm/Group | SHAPE Measurement
Started | 21 (Only subjects with portal hypertension in "overall study" were eligible to progress to "follow-up")
Completed | 11
Not Completed | 10
Not completed — Lost to Follow-up | 10

BASELINE CHARACTERISTICS:
Arm/Group | SHAPE Measurement
Number analyzed (Participants) | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 121
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 41
  White | 79
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 125

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Accuracy of SHAPE Liver Pressure Estimates (in dB) for Diagnosing Portal Hypertension With Catheter Pressure Measurements (in mmHg) as the Reference Standard
Description: Evaluate the use of in vivo subharmonic aided pressure estimation (SHAPE as the difference between the optimized subharmonic signal in a hepatic vein and in the portal vein) as a first quantitative screening modality for determining the presence of clinically significant portal hypertension in patients undergoing a transjugular liver biopsy compared to catheter based hepatic-venous pressure gradient measurements (HVPG in mmHg as the reference standard).
Time Frame: up to 1 day
Measure: Number; unit: diagnostic accuracy in percent
Arm/Group | SHAPE Measurement
Number analyzed (Participants) | 113
diagnostic accuracy in percent | 95

2. Primary Outcome: SHAPE Liver Pressure Estimates (in dB) Correlation With Catheter Pressure Measurements (in mmHg)
Description: Evaluate the correlation between in vivo subharmonic aided pressure estimation (SHAPE as the difference between the optimized subharmonic signal in a hepatic vein and catheter based hepatic-venous pressure gradient measurements (HVPG in mmHg) in patients undergoing a transjugular liver biopsy.
Time Frame: up to 1 day
Measure: Number; unit: correlation coefficient
Arm/Group | SHAPE Measurement
Number analyzed (Participants) | 113
correlation coefficient | 0.68

3. Primary Outcome: Comparing SHAPE Results With Blood Work and Concomitant Imaging in Portal Hypertension Patients
Description: Determine if SHAPE measurements (in dB) can provide a quantitative, noninvasive measurement of hepatic venous pressure gradient (HVPG) to monitor disease progression or treatment response in patients identified with portal hypertension by comparing the results to repeat biopsies and/or clinical outcomes.
Time Frame: up to 2 hours
Population: Only subjects with clinically significant portal hypertension were included in the follow-up study
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | SHAPE Measurement
Number analyzed (Participants) | 11
dB
  SHAPE values in responders: number analyzed (Participants) | 10
  SHAPE values in responders | -4.01 (3.61)
  SHAPE value in non-responders: number analyzed (Participants) | 1
  SHAPE value in non-responders | 2.33 (0)

ADVERSE EVENTS:
Time Frame: 2 hours after infusion of the ultrasound contrast agent
Arm/Group | SHAPE Measurement
All-Cause Mortality (participants affected / at risk) | 0/125
Serious Adverse Events (participants affected / at risk) | 0/125
Other Adverse Events (participants affected / at risk) | 0/125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-21): https://cdn.clinicaltrials.gov/large-docs/45/NCT02489045/Prot_SAP_000.pdf